CLINICAL TRIAL: NCT04452344
Title: Opioid Analgesic Reduction Study (OARS): Managing Acute Post-Operative Surgical Pain
Brief Title: Opioid Analgesic Reduction Study
Acronym: OARS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); University of Rochester (Other); University of Maryland, Baltimore (Other); University of Illinois at Chicago (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Cecile A. Feldman, DMD, Dean and Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Pro2020002299; 5UH3DE028860-05 (NIH)
Record Dates: First submitted 2020-04-07; First posted 2020-06-30 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use
Keywords: 3rd molar extraction pain model; Opioid Analgesics; Opioid Diversion; Over the counter analgesics; Acetaminophen; Ibuprofen; Hydrocodone; Opioid Addiction; Pain Management; Satisfaction
MeSH Terms: conditions — Opioid-Related Disorders; Agnosia; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was a double-blinded study. The participant, care provider, site directors and site research coordinators were all blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid (Active Comparator): Combination analgesic of hydrocodone 5mg/acetaminophen 300 mg and a placebo pill.
  Interventions: Drug: opioid-containing analgesic
- Non-Opioid (Active Comparator): Combination of ibuprofen 400 mg/acetaminophen 500 mg
  Interventions: Drug: two over-the-counter analgesics

INTERVENTIONS:
Drug: opioid-containing analgesic — hydrocodone/ acetaminophen combination product
  Arms: Opioid
Drug: two over-the-counter analgesics — combination of over-the-counter analgesics (ibuprofen/acetaminophen)
  Arms: Non-Opioid

SUMMARY:
The goal is to provide health care professionals, including dentists, with the best possible evidence for clinical decision making when deciding upon analgesics for acute post-surgical pain management, a double-blind, stratified randomized clinical trial will be conducted to test the hypothesis that a combination of over-the-counter non-opioid containing analgesics is at least as, if not more, effective (non-inferior) than the most commonly prescribed opioid analgesic. The impacted 3rd molar extraction model will be used due to the predictable severity of the post-operative pain and generalizability of results.

This double-blind, prospective, stratified, randomized pragmatic clinical trial will use the impacted 3rd molar extraction pain model.

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all of the following criteria to be eligible to participate in the study:

* Be able to understand the informed consent.
* Provide signed and dated informed consent form
* Be able to understand all directions for data gathering instruments in English
* Be willing and able to comply with all study procedures and be available for the duration of the study
* Planning to undergo extraction of one or more partial or fully impacted mandibular 3rd molars
* Be 18 years or older
* Be in good general health as evidenced by medical history
* Women must agree to use one of the following methods of contraception while participating in this study:

  * contraceptive pill
  * intra-uterine device
  * condoms
  * abstinence

Exclusion Criteria:

Participants who self-report the following history will be excluded from participating:

* History of gastrointestinal bleeding and/or peptic ulcer
* History of renal disease (excluding kidney stones)
* History of hepatic disease
* History of bleeding disorder
* History of respiratory depression
* Any prior respiratory effect of an opioid or other anesthetic drugs that required respiratory support postoperatively
* Active or untreated asthma
* History of known allegoric reaction to ibuprofen, acetaminophen, hydrocodone, and/or anesthesia
* Currently taking any of the following medications:

  * CYP3A4 inhibitor, such as macrolide antibiotics (e.g., erythromycin), azole-antifungal agents (e.g., ketoconazole), and protease inhibitors (e.g., ritonavir), which may increase plasma concentrations of hydrocodone bitartrate and acetaminophen and prolong opioid adverse reactions, and which may cause potentially fatal respiratory depression
  * CNS depressants.
* Consumes 3 or more alcoholic drinks every day and/or has a history of alcoholism
* History of drug or alcohol abuse
* Family history of drug or alcohol abuse in a first-degree relative
* Has had no more than one opioid prescription filled within the past 12 months
* Currently pregnant or lactating

Participants would also be excluded due to any additional criteria that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study which includes:

* Prior participation in this study
* Inability or refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1815 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Feldman, DMD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (5):
- United States (5):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Rutgers School of Dental Medicine, Newark, New Jersey
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
Electronic Data Capture (EDC) will be used extensively throughout the course of the study for the collection of patient data as well as driving operational/logistical workflows. The database with data dictionary will be available.
Time Frame: 12 months after publication
Access Criteria: Request data access from the PI.

REFERENCES:
- [Derived] Feldman CA, Fredericks-Younger J, Desjardins PJ, Malmstrom H, Miloro M, Warburton G, Ward BB, Ziccardi VB, Greenberg P, Andrews T, Matheson PB, Benoliel R, Fine DH, Lu SE. Nonopioid vs opioid analgesics after impacted third-molar extractions: The Opioid Analgesic Reduction Study randomized clinical trial. J Am Dent Assoc. 2025 Feb;156(2):110-123.e9. doi: 10.1016/j.adaj.2024.10.014. Epub 2025 Jan 4. PMID 39755971
- [Derived] Feldman CA, Fredericks-Younger J, Lu SE, Desjardins PJ, Malmstrom H, Miloro M, Warburton G, Ward B, Ziccardi V, Fine D. The Opioid Analgesic Reduction Study (OARS)-a comparison of opioid vs. non-opioid combination analgesics for management of post-surgical pain: a double-blind randomized clinical trial. Trials. 2022 Feb 17;23(1):160. doi: 10.1186/s13063-022-06064-8. PMID 35177108

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Opioid | Opioid
Started | 909 | 906
Completed | 897 | 889
Not Completed | 12 | 17
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — No Post-Op Visit | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Opioid | Opioid | Total
Number analyzed (Participants) | 909 | 906 | 1815
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 25.58 (5.97) | 25.81 (6.50) | 25.69 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 457 | 453 | 910
  Male | 452 | 453 | 905
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 279 | 282 | 561
  Non-Hispanic Asian | 141 | 131 | 272
  Non-Hispanic Black | 255 | 257 | 512
  Non-Hispanic White | 179 | 178 | 357
  Other | 32 | 30 | 62
  Did Not Want to Report | 23 | 28 | 51
3rd molars extracted [Mean (Standard Deviation); unit: teeth] — Number of 3rd molars extracted (range = 1 to 4)
  teeth | 2.75 (1.17) | 2.75 (1.21) | 2.75 (1.19)
Impacted full bony 3rd molars extracted [Mean (Standard Deviation); unit: teeth] — Number of full bony impacted 3rd molars extracted (range=0 to 4)
  teeth | .96 (1.23) | 0.98 (1.22) | .97 (1.23)

OUTCOME MEASURES:

1. Primary Outcome: Composite Pain 1
Description: Before going to sleep participants are asked to rate their "worst pain experienced", "least pain experienced" and "average pain experienced" during the day along with "pain now." Upon waking participants were asked to rate their "worst pain experienced", "least pain experienced" and "average pain experienced" during the night along with "pain now." A NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine was used. Composite Pain 1 is the average of all ratings provided at the end of day of surgery (day 1) and when waking up the next morning (1 night after surgery).
Time Frame: End of day of surgery (day 1) and when waking up the next morning (1 night after surgery)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
units on a scale | 3.77 [3.58 to 3.96] | 4.47 [4.28 to 4.65]

2. Primary Outcome: Composite Pain 2
Description: Before going to sleep participants are asked to rate their "worst pain experienced", "least pain experienced" and "average pain experienced" during the day along with "pain now." Upon waking participants were asked to rate their "worst pain experienced", "least pain experienced" and "average pain experienced" during the night along with "pain now." A NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine was used. Composite Pain 2 is the average of all ratings provided day after surgery (day 2) and when waking up the next morning (2nd night after surgery).
Time Frame: End of day of the second day after surgery (day 2) and when waking up the next morning (2nd night after surgery)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
units on a scale | 3.20 [3.01 to 3.39] | 3.48 [3.29 to 3.67]

3. Primary Outcome: Composite Pain 3
Description: Before going to sleep participants are asked to rate their "worst pain experienced", "least pain experienced" and "average pain experienced" during the day along with "pain now." Upon waking participants were asked to rate their "worst pain experienced", "least pain experienced" and "average pain experienced" during the night along with "pain now." A NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine was used. Composite Pain 3 is the average of all ratings provided two days after surgery (day 3) and when waking up the 3rd morning after surgery (3rd night after surgery).
Time Frame: End of day of the third day after surgery (day 3) and when waking up the next morning (3rd night after surgery)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
units on a scale | 2.97 [2.78 to 3.16] | 3.06 [2.87 to 3.25]

4. Primary Outcome: Composite Pain All
Description: Before going to sleep participants are asked to rate their "worst pain experienced", "least pain experienced" and "average pain experienced" during the day along with "pain now." Upon waking participants were asked to rate their "worst pain experienced", "least pain experienced" and "average pain experienced" during the night along with "pain now." A NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine was used. Composite Pain All is the average of the ratings provided at the end of first 7 days after surgery (days 1 thru 7) and when waking up the first 7 mornings (1st thru 7th nights after surgery).
Time Frame: End of first 7 days after surgery (days 1 thru 7) and when waking up the first 7 mornings (1st thru 7th nights after surgery)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
units on a scale | 2.73 [2.54 to 2.92] | 2.94 [2.74 to 3.13]

5. Primary Outcome: Overall Satisfaction
Description: Participant rating on a five point Likert Scale (1=very satisfied, 2=satisfied, 3=neither satisfied or dissatisfied, 4=dissatisfied, 5=very dissatisfied) to the question: "Overall, how satisfied were you with your current pain medication?"
Time Frame: At time of post-operative visit (day 9 +/- 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
Participants
  Very Satisfied | 355 | 308
  Satisfied | 409 | 395
  Neither satisfied nor dissatisfied | 87 | 122
  Dissatisfied | 33 | 54
  Very dissatisfied | 12 | 12
  MIssing | 13 | 15

6. Primary Outcome: Pain Worst 1
Description: Participants are asked to rate the worst pain they experienced during the day (recorded before going to sleep) and overnight (recorded when waking up) on a NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine. Pain Worst 1 is the average of the ratings provided at the end of day of surgery (day 1) and when waking up the next morning (1 night after surgery).
Time Frame: End of day of surgery (day 1) and when waking up the next morning (1 night after surgery)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 4.90 [4.59 to 5.21] | 5.79 [5.47 to 6.10]

7. Primary Outcome: Pain Worst 2
Description: Participants are asked to rate the worst pain they experienced during the day (recorded before going to sleep) and overnight (recorded when waking up) on a NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine. Pain Worst 2 is the average of the ratings provided at the end of day of after surgery (day 2) and when waking up the next morning (2nd night after surgery.)
Time Frame: End of day of after surgery (day 2) and when waking up the next morning (2nd night after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 4.17 [3.86 to 4.48] | 4.48 [4.17 to 4.80]

8. Primary Outcome: Pain Worst 3
Description: Participants are asked to rate the worst pain they experienced during the day (recorded before going to sleep) and overnight (recorded when waking up) on a NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine. Pain Worst 3 is the average of the ratings provided at the end of 2nd day of after surgery (day 3) and when waking up the next morning (3rd night after surgery).
Time Frame: End of 2nd day of after surgery (day 3) and when waking up the next morning (3rd night after surgery)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 3.97 [3.65 to 4.28] | 3.96 [3.65 to 4.27]

9. Primary Outcome: Pain Worst All
Description: Participants are asked to rate the worst pain they experienced during the day (recorded before going to sleep) and overnight (recorded when waking up) on a NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine. Pain Worst all is the average of the ratings provided at the end of first 7 days after surgery (days 1 thru 7) and when waking up the first 7 mornings (1st thru 7th nights after surgery).
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 3.66 [3.34 to 3.97] | 3.79 [3.48 to 4.11]

10. Primary Outcome: Pain Average 1
Description: Participants are asked to rate the average pain they experienced during the day (recorded before going to sleep) and overnight (recorded when waking up) on a NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine. Pain Average 1 is the average of the ratings provided at the end of day of surgery (day 1) and when waking up the next morning (1 night after surgery)
Time Frame: End of day of surgery (day 1) and when waking up the next morning (1 night after surgery)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 3.75 [3.57 to 3.94] | 4.47 [4.29 to 4.66]

11. Primary Outcome: Pain Average 2
Description: Participants are asked to rate the average pain they experienced during the day (recorded before going to sleep) and overnight (recorded when waking up) on a NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine. Pain Average 2 is the average of the ratings provided at the end of day of after surgery (day 2) and when waking up the next morning (2nd night after surgery.)
Time Frame: End of day of after surgery (day 2) and when waking up the next morning (2nd night after surgery)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 3.18 [3.00 to 3.37] | 3.49 [3.31 to 3.68]

12. Primary Outcome: Pain Average 3
Description: Participants are asked to rate the average pain they experienced during the day (recorded before going to sleep) and overnight (recorded when waking up) on a NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine. Pain Average 3 is the average of the ratings provided at the end of 2nd day of after surgery (day 3) and when waking up the next morning (3rd night after surgery).
Time Frame: End of 2nd day of after surgery (day 3) and when waking up the next morning (3rd night after surgery)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 2.97 [2.78 to 3.15] | 3.07 [2.89 to 3.26]

13. Primary Outcome: Pain Average All
Description: Participants are asked to rate the average pain they experienced during the day (recorded before going to sleep) and overnight (recorded when waking up) on a NRS scale of 0 to 10 where 0=no pain and 10=pain as bad as you can imagine. Pain Average all is the average of the ratings provided at the end of first 7 days after surgery (days 1 thru 7) and when waking up the first 7 mornings (1st thru 7th nights after surgery).
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 2.69 [2.50 to 2.88] | 2.95 [2.76 to 3.14]

14. Secondary Outcome: Number of Participants Receiving Rescue Medication
Description: Participant receiving additional pain medication (oxycodone) as study analgesic is not managing pain sufficiently
Time Frame: At post operative visit (9 days after surgery +/- 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
Participants | 26 | 54

15. Secondary Outcome: Pain Interference 1
Description: Participants were asked to rate, on a 5 point Likert Scale, how much did pain interfered with their day to day activities, work around the home, ability to participate in social activities, enjoyment of life, the things you usually do for fun, enjoyment of social activities, household chores, family life, your ability to concentrate, enjoyment of recreational activities, tasks away from home {scale: 1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit, 5=very much} and How often did pain keep you from socializing with others? {scale=1=never, 2=rarely, 3=sometimes, 4=often, 5=always} Pain Interference 1 is the average ratings provided at the end of the day of surgery. Lower scores are better.
Time Frame: End of the day of surgery (day 1)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 2.75 [2.65 to 2.85] | 3.11 [3.01 to 3.21]

16. Secondary Outcome: Pain Interference 2
Description: Participants were asked to rate, on a 5 point Likert Scale, how much did pain interfered with their day to day activities, work around the home, ability to participate in social activities, enjoyment of life, the things you usually do for fun, enjoyment of social activities, household chores, family life, your ability to concentrate, enjoyment of recreational activities, tasks away from home {scale: 1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit, 5=very much} and How often did pain keep you from socializing with others? {scale=1=never, 2=rarely, 3=sometimes, 4=often, 5=always} Pain Interference 2 is the average ratings provided at the end of day after surgery (day 2). Lower scores are better.
Time Frame: End of the first full day after surgery (day 2)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 2.27 [2.17 to 2.37] | 2.50 [2.40 to 2.59]

17. Secondary Outcome: Pain Interference 3
Description: Participants were asked to rate, on a 5 point Likert Scale, how much did pain interfered with their day to day activities, work around the home, ability to participate in social activities, enjoyment of life, the things you usually do for fun, enjoyment of social activities, household chores, family life, your ability to concentrate, enjoyment of recreational activities, tasks away from home {scale: 1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit, 5=very much} and How often did pain keep you from socializing with others? {scale=1=never, 2=rarely, 3=sometimes, 4=often, 5=always} Pain Interference 3 is the average ratings provided at the end of 2nd day after surgery (day 3). Lower scores are better.
Time Frame: End of the second full day after surgery (day 3)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 2.20 [2.10 to 2.30] | 2.34 [2.24 to 2.44]

18. Secondary Outcome: Pain Interference All
Description: Participants were asked to rate, on a 5 point Likert Scale, how much did pain interfered with their day to day activities, work around the home, ability to participate in social activities, enjoyment of life, the things you usually do for fun, enjoyment of social activities, household chores, family life, your ability to concentrate, enjoyment of recreational activities, tasks away from home {scale: 1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit, 5=very much} and How often did pain keep you from socializing with others? {scale=1=never, 2=rarely, 3=sometimes, 4=often, 5=always} Pain Interference ALL is the average ratings provided at the end of the 1st seven days after surgery (days 1 thru 7). Lower scores are better.
Time Frame: First 7 days after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 2.09 [2.01 to 2.18] | 2.21 [2.13 to 2.30]

19. Secondary Outcome: Sleep 1
Description: Participants were asked to rate the overall quality of their sleep the 1st night after surgery on a NRS scale of 0 to 10 where 0=excellent and 10=very poor. Sleep 1 is the rating provided when first waking up the day after surgery.
Time Frame: When first waking up the day after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 4.28 [4.02 to 4.54] | 4.62 [4.36 to 4.88]

20. Secondary Outcome: Sleep 2
Description: Participants were asked to rate the overall quality of their sleep the 2nd night after surgery on a NRS scale of 0 to 10 where 0=excellent and 10=very poor. Sleep 2 is the rating provided when first waking up the second day after surgery.
Time Frame: When first waking up the 2nd day after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 4.10 [3.84 to 4.35] | 4.14 [3.88 to 4.40]

21. Secondary Outcome: Sleep 3
Description: Participants were asked to rate the overall quality of their sleep the 3rd night after surgery on a NRS scale of 0 to 10 where 0=excellent and 10=very poor. Sleep 1 is the rating provided when first waking up the third day after surgery.
Time Frame: When first waking up the 3rd day after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 3.78 [3.52 to 4.04] | 3.82 [3.56 to 4.08]

22. Secondary Outcome: Sleep All
Description: Participants were asked to rate the overall quality of their sleep for the first 7 nights after surgery on a NRS scale of 0 to 10 where 0=excellent and 10=very poor. Sleep All is the average rating provided for all seven nights.
Time Frame: First 7 nights after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 909 | 906
score on a scale | 3.69 [3.44 to 3.94] | 3.62 [3.37 to 3.87]

23. Secondary Outcome: Potential for Opioid Tablet Diversion
Description: Number of returned opioid analgesic capsules at post operative visit (9 days after surgery +/- 5 days)
Time Frame: At post operative visit (9 days after surgery +/- 5 days)
Measure: Mean (95% Confidence Interval); unit: capsules
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 896 | 891
capsules | 0 [0 to 0] | 8.55 [7.50 to 9.60]

24. Post Hoc Outcome: Satisfaction 1
Description: Participants were asked "overall, how satisfied were you with your current pain medication". Responses were provided on a five point Likert Scale (1=very satisfied, 2=satisfied, 3=neither satisfied or dissatisfied, 4=dissatisfied, 5=very dissatisfied) Satisfaction 1 is the average of the response provided for the day of surgery and the 1st night after surgery.
Time Frame: Day of surgery (day 1) and 1 night after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 386 | 388
score on a scale | 2.22 [2.13 to 2.30] | 2.38 [2.30 to 2.47]

25. Post Hoc Outcome: Satisfaction 2
Description: Participants were asked "overall, how satisfied were you with your current pain medication". Responses were provided on a five point Likert Scale (1=very satisfied, 2=satisfied, 3=neither satisfied or dissatisfied, 4=dissatisfied, 5=very dissatisfied) Satisfaction 2 is the average of the response provided for the 1st day of after surgery (day 2) and the 2nd night after surgery.
Time Frame: Day after surgery (day 2) and 2nd night after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 386 | 388
score on a scale | 2.17 [2.08 to 2.26] | 2.27 [2.18 to 2.35]

26. Post Hoc Outcome: Satisfaction 3
Description: Participants were asked "overall, how satisfied were you with your current pain medication". Responses were provided on a five point Likert Scale (1=very satisfied, 2=satisfied, 3=neither satisfied or dissatisfied, 4=dissatisfied, 5=very dissatisfied) Satisfaction 3 is the average of the response provided for the 2nd day of after surgery (day 3) and the 3nd night after surgery.
Time Frame: Second day after (day 3) and third night after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 386 | 388
score on a scale | 2.21 [2.12 to 2.30] | 2.30 [2.21 to 2.39]

27. Post Hoc Outcome: Satisfaction All
Description: Participants were asked "overall, how satisfied were you with your current pain medication". Responses were provided on a five point Likert Scale (1=very satisfied, 2=satisfied, 3=neither satisfied or dissatisfied, 4=dissatisfied, 5=very dissatisfied) Satisfaction ALL is the average of the ratings provided at the end of first 7 days after surgery (days 1 thru 7) and when waking up the first 7 mornings (1st thru 7th nights after surgery).
Time Frame: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Opioid | Opioid
Number analyzed (Participants) | 386 | 388
score on a scale | 2.24 [2.14 to 2.34] | 2.27 [2.18 to 2.36]

ADVERSE EVENTS:
Time Frame: Adverse even data was collected between the time of surgery and the post-operative visit which was 9 days +/- 5 days.
Arm/Group | Non-Opioid | Opioid
All-Cause Mortality (participants affected / at risk) | 0/909 | 0/906
Serious Adverse Events (participants affected / at risk) | 1/909 | 2/906
Other Adverse Events (participants affected / at risk) | 58/909 | 51/906
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Opioid (N=909) | Opioid (N=906)
Spider Bite (Infections and infestations) | 0 (0) | 1 (1) — Patient hospitalized due to complications from a spider bite
Infection & Swelling (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Opioid (N=909) | Opioid (N=906)
Pain (Nervous system disorders) | 25 (25) | 27 (27)
Bleeding (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Skin rash (Immune system disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Other (General disorders) | 20 (20) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT04452344/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04452344/ICF_000.pdf